CLINICAL TRIAL: NCT07195604
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Dose of HRS-2162 Injection in Healthy Subjects
Brief Title: A Single Ascending Dose of HRS-2162 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-2162-101
Record Dates: First submitted 2025-09-14; First posted 2025-09-26 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Reversal of Neuromuscular Blockade

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Dose Level：A1(Part1) (Experimental): Subject will receive HRS-2162 at dose level A1. Subject will receive placebo at dose level A1.
  Interventions: Drug: HRS-2162; Drug: Placebo
- Dose Level：A2(Part1) . (Experimental): Subject will receive HRS-2162 at dose level A2. Subject will receive placebo at dose level A2.
  Interventions: Drug: HRS-2162; Drug: Placebo
- Dose Level：B(Part1+Part2) (Experimental): Subject will receive HRS-2162 at dose level B. Subject will receive placebo at dose level B.
  Interventions: Drug: HRS-2162; Drug: Placebo
- Dose Level：C(Part1) (Experimental): Subject will receive HRS-2162 at dose level C. Subject will receive placebo at dose level C.
  Interventions: Drug: HRS-2162; Drug: Placebo
- Dose Level：D(Part1+Part3) (Experimental): Subject will receive HRS-2162 at dose level D. Subject will receive placebo at dose level D.
  Interventions: Drug: HRS-2162; Drug: Placebo
- Dose Level：E(Part1) (Experimental): Subject will receive HRS-2162 at dose level E. Subject will receive placebo at dose level E.
  Interventions: Drug: HRS-2162; Drug: Placebo
- Dose Level：F(Part3) (Experimental): Subject will receive HRS-2162 at dose level F
  Interventions: Drug: HRS-2162

INTERVENTIONS:
Drug: HRS-2162 — HRS-2162
Drug: Placebo — Placebo
  Arms: Dose Level：A1(Part1); Dose Level：A2(Part1) .; Dose Level：B(Part1+Part2); Dose Level：C(Part1); Dose Level：D(Part1+Part3); Dose Level：E(Part1)

SUMMARY:
The study is being conducted to evaluate the safety and tolerability of HRS-2162 injection in a single dose in healthy subjects, as well as the characteristics of PK/PD

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily signed the informed consent form.
2. Applicants must be between 18 and 45 years old at the time of signing the informed consent form, and both men and women are eligible .
3. ASA classification is Grade I (only Parts Two and three)
4. Male weight ≥50 kg, female weight ≥45 kg, body mass index between 19 and 28 kg/m ².
5. Adopt efficient contraceptive measures

Exclusion Criteria:

1. Those with a past or current clinical acute or chronic disease
2. Those with a history of hereditary bleeding or coagulation disorders or non-traumatic bleeding .
3. Those with a history of neuromuscular diseases or poliomyelitis
4. Those with a history of anesthesia complications.
5. Those whose laboratory test results during the screening period or baseline period exceed the normal range and have clinical significance
6. The blood pressure of the subjects was abnormal and was judged by the researchers to be of clinical significance
7. The subject has a history of severe systemic allergies for any reason.
8. The subjects took steroid hormone drugs within 7 half-lives or 14 days before administrationSmoke ≥5 cigarettes per day within 3 months prior to the study.
9. History of drug abuse.
10. Those who the researchers considered unsuitable for inclusion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | From ICF signing date to Day7

SECONDARY OUTCOMES:
Maximum observed concentration of HRS-2162 (Cmax) | 0 hour to 24 hour after administration
Area under the serum concentration time curve (AUC) of HRS-2162 | 0 hour to 24 hour after administration
Time to maximum observed concentration (Tmax) of HRS-2162 | 0 hour to 24 hour after administration
Half-life (T1/2) of HRS-2162 | 0 hour to 24 hour after administration
Clearance (CL) of HRS-2162 | 0 hour to 24 hour after administration
Volume of distribution (Vz) of HRS-2162 | 0 hour to 24 hour after administration
Efficacy endpoint: The time required from the administration of the investigational drug to the recovery of the TOFr value (T4/T1 value) | 0 hour to 1 hour after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Academy of Medical Sciences &Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided